CLINICAL TRIAL: NCT02565524
Title: Exploration and Characterization of the Phenotypic and Genetic Profile of Patients With Early Onset Schizophrenia Associated With Autism Spectrum Disorder and Their First-degree Relatives (GenAuDiss).
Brief Title: the Phenotypic and Genetic Profile of Patients With Early Onset Schizophrenia Associated With Autism Spectrum Disorder.
Acronym: GenAuDiss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-HPNCL08
Record Dates: First submitted 2015-07-29; First posted 2015-10-01 (Estimated); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Schizophrenia; Dissociative Disorders
Keywords: schizophrenia; early dissociative disorder; genetic
MeSH Terms: conditions — Schizophrenia; Dissociative Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- genetic and phenotypic profile (Experimental): blood sample, clinical and neurocognitive assessment
  Interventions: Other: genetic and phenotypic profile

INTERVENTIONS:
Other: genetic and phenotypic profile — Genetic and phenotypic profile, clinical and neurocognitive assessment for child with Schizophrenia and autism, their parents and brotherhood

SUMMARY:
Early onset schizophrenia "early dissociative disorder" is a rare disorder with a low incidence of approximately (1/5000 to 1/20000). Its link with autism spectrum disorders remains unknown although both are serious neurodevelopmental diseases. As part of the 2011-2013 Interregional hospital Clinical Research program, University Department of Child and Adolescent Psychiatry Pediatric Hospitals of CHU de Nice Lenval identified patients with a complex phenotype characterized by an early schizophrenia associated with autism spectrum disorders and developmental disabilities in mild to moderate. This phenotype could be a new syndrome.

The goal of our project is to define the genetic causes of this phenotype. The technique of high throughput sequencing will be used to obtain the sequence of exomes of these patients and their families. This study will therefore be important to give an accurate diagnosis for patients and their families. Moreover, we believe that this project will identify new genes involved allowing a better understanding of the pathophysiology. Recent studies show the involvement of mutations in several genes (eg NRXN1 and UPF3B) in these different clinical phenotypes. However, the genetic basis of the childhood and early onset schizophrenia are much less well known than those of autism spectrum disorder

DETAILED DESCRIPTION:
Introduction: Early-onset Schizophrenia (EOS) is a rare and severe condition displaying early dissociative disorder (i.e., age of onset < 18 years). A higher rate of neurodevelopmental abnormalities is observed in EOS compared to adult onset schizophrenia (AOS). Thus, patients affected by EOS typically present intellectual, learning, communication or neuromotor impairments, as well as attention deficit hyperactivity disorder. Early signs of autism spectrum disorders (ASD) are also found in 30% of patients with EOS.

Cytogenetics abnormalities, including copy number variations (CNVs), are frequent in neurodevelopmental disorders and have been linked to ASD physiopathology. Implicated genes encode proteins playing a role in brain development, synaptic morphology, plasticity and neurogenesis. In addition, an increasing number of genetic abnormalities are shared by EOS and ASD, suggesting that schizophrenia can be considered a neurodevelopmental disorder.

The main objective of the present study is to identify mutations in genes involved in neurodevelopmental pathways in our cohort of patients affected by both EOS and ASD.

Method and analysis: We describe here a multicenter study in a pediatric population named "Exploration and characterization of genetic and phenotypic profile of the 'early dissociative disorder' associated with autism spectrum disorder (GenAuDiss)". The study started in April 2014. The inclusion criteria are: age 7 to 22 years, diagnoses of EOS with co-morbid ASD and IQ > 50; as well as parents and siblings of the included patients.

We perform standardized psychiatric assessments (MINI, K-SADS-PL, PANSS, SANS, TCI 226, and AQ) and neurocognitive evaluations (IQ, TMT A/B, and verbal fluency). Then, we study variants of the coding part of the DNA (exome), using next generation sequencing (NGS) process on trio (mother, father, and child). Divers bio-informatics tools such as RVIS and PolyPhen-2 will be used to prioritize the potential candidate genes. The inclusion period of this study will end in November 2019.

Ethics and dissemination: The study protocol was approved by the Ethics Committee 'Sud Méditerrané V' (number 14.002) and by the French National Agency for Medicines and Health Products Safety (ANSM 2013-A01699-36). All patients, their parents and siblings signed informed consent upon enrolment in the study.

Results of the present study should help to unravel the molecular pathology of EOS, paving the way for an early therapeutic intervention

ELIGIBILITY:
Inclusion Criteria:

Of the child:

* ≥ 7 years, <18 (below 7 years the diagnosis of schizophrenia is not possible)
* Schizophrenia Diagnosis done using the diagnostic tool Kiddie sads
* Autism Diagnosis done using the diagnostic scale Autism Diagnostic interview (ADI-R)
* Intelligence quotient (IQ) ≥ 50 at Wechsler Intelligence Scale for Children (WISC) IV abridged version
* Clinical examination
* Affiliation to social security
* Obtaining the authorization of the holders of parental authority

Brothers and sisters:

* Minor or Major
* Similarly biological parents
* Clinical examination
* Affiliation to social security
* Obtaining the authorization of the holders of parental authority for minors or informed consent for major

Parents:

* Biological Parent
* Clinical examination
* Affiliation to social security
* Informed Consent

Exclusion Criteria:

Of the child:

* Children refusing to participate
* Children without verbal language

Brothers and sisters:

* Children refusing to participate
* Adults protected by law

Parents:

* Refusing to participate
* Adults are protected by law

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 111 (Actual)
Dates: Start 2014-05-18 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
characterization of the genetic abnormalities associated to Early Onset Schizophrenia phenotypes by performing standard karyotype | inclusion visit
  A standard karyotype at a resolution of 300 to 400 bands per haploid lot. It can diagnose numerical anomalies and certain structural abnormalities such as reciprocal translocations, inversions, deletions.
  A standard karyotype at a resolution of 300 to 400 bands per haploid lot is established initially. It can diagnose numerical anomalies and certain structural abnormalities such as reciprocal translocations, inversions, deletions Big.
  The pathological nature of these mutations will be stutied on the gene function and reaches its pattern of expression.
characterization of the genetic abnormalities associated to Early Onset Schizophrenia phenotypes by performing search CGG | inclusion visit
  A search of the CGG expansion hypermethylated in the 5 'UTR of the FMR1 gene mutation that causes Fragile X syndrome.
characterization of the genetic abnormalities associated to Early Onset Schizophrenia phenotypes by performing whole exome sequencing | inclusion visit
  Whole Exome Sequencing on trio (mother, father and child); This technology has demonstrated its power in recent years to determine the genetic causes of many rare diseases (Ropers, HH., 2012).

SECONDARY OUTCOMES:
Intensity of positive symptoms of schizophrenia | inclusion visit
  Evaluation of the intensity of positive and negative symptoms, general psychopathology and subtypes of schizophrenia by using positive and negative syndrome scale (PANSS)
Co-morbid psychiatric diagnosis | inclusion visit
  Evaluation of clinical profile: by using K-SADS-PL scale for DSM IV-TR / DSM-5 co-morbid psychiatric diagnosis of patients and minor siblings and by using MINI assessments for DSM IV-TR / DSM 5 psychiatric diagnosis of parents and major siblings.
Evaluation of executive and attentional by the verbal fluency test | inclusion visit
  Evaluation of executive and attentional functions of patients using Trail Making Test (TMT) A and B and verbal fluency;
Clinical evaluation of autistic symptoms | inclusion visit
  Clinical evaluation of autistic symptoms by using AQ (Baron-Cohen) in siblings and parents
Neurocognitive profile | inclusion visit
  Evaluation of cognitive functioning by Wechsler Intelligence Scale for Children Scale IV (WISC IV).full version in patient and WISC IV abridged version in minor siblings; Wechsler Adult Intelligence Scale-III (WAIS III) in a short form in adult siblings and parents
Personality dimensional test | inclusion visit
  Personality dimensional test using computerized version of TCI 226 (Cloninger) in parents

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle DOR, MD, Principal Investigator — Fondation Lenval
Locations (1):
- Fondation Lenval, Nice, France

REFERENCES:
- [Derived] Fernandez A, Dor E, Maurin T, Laure G, Menard ML, Drozd M, Poinso F, Bardoni B, Askenazy F, Thummler S. Exploration and characterisation of the phenotypic and genetic profiles of patients with early onset schizophrenia associated with autism spectrum disorder and their first-degree relatives: a French multicentre case series study protocol (GenAuDiss). BMJ Open. 2018 Jul 5;8(7):e023330. doi: 10.1136/bmjopen-2018-023330. PMID 29980548